CLINICAL TRIAL: NCT01104194
Title: The Effects of Omega-3 Fatty Acids Dietary Supplements (Fish-oil) on Mood and Cognitive Functions of Healthy Individuals
Brief Title: Effects of Fish-oil on Mood and Cognitive Functions of Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Prof AJW Van der Does, Leiden University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P07.063
Record Dates: First submitted 2010-04-12; First posted 2010-04-15 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-07

CONDITIONS: Depression
Keywords: depression; cognition; heart rate variability; omega-3 fatty acids; Depression (in remission) (vulnerability to depression)
MeSH Terms: conditions — Depression | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fish-oil (Experimental)
  Interventions: Dietary Supplement: omega-3 fatty acids supplements (fish oil)
- Placebo (Placebo Comparator): Olive oil capsules, identical in appearance to fish oil capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acids supplements (fish oil) — 1.74g eicosapentaenoic acid (EPA) and 0.25g docosahexaenoic acid (DHA)
  Arms: Fish-oil
Dietary Supplement: Placebo — softgel capsules (identical in appearance to fish oil capsules) containing olive oil. 3 capsules/day, 4 weeks
  Arms: Placebo

SUMMARY:
The investigators recently found a positive effect of omega-3 supplements on cognitive function in healthy individuals after 4 weeks (J of Psychopharmacology 2009, 23: 831-840). The investigators hypothesize that 4 weeks consumption of omega-3 supplements in previously depressed individuals will positively affect their cognitive functions.

Secondly, low Heart Rate Variability (HRV) is a risk factor for cardiovascular disease. Some studies have found low HRV in patients with depression. No studies have investigated the effects of omega-3 fatty acid supplements on Heart Rate Variability in individuals with a history of depression. The investigators will test the hypotheses that omega-3 supplements lead to an improvement of heart rate variability indices in healthy volunteers with a history of depression.

ELIGIBILITY:
Inclusion Criteria:

* Dutch-speaking men and women
* Normal weight (BMI between 18 and 27).
* Regular diets, not containing fish more than once a week.
* History of depression (at least one major depressive episode in the past).

Exclusion Criteria:

* Currently more than mildly depressed (BDI-II-NL score higher than 19, or score on the suicidality item of this scale higher than 1).
* Current or past psychosis
* Current substance abuse or past substance dependence
* Smoking or current use of soft drugs (current = month prior to study till completion)
* Any hard drug use (lifetime)
* More than 3 alcoholic consumptions/day

Participants will be asked to keep their dietary habits constant throughout the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Cognition | 4 weeks
  Battery of test measuring emotional and neutral information processing. Largest effect expected on Decision Making Test (cf. Antypa et al., 2009) and Emotion Recognition Test.
Heart Rate Variability | 4 weeks

SECONDARY OUTCOMES:
Mood states | 4 weeks
  Fatigue, Anger, Tension, Anxiety, Vigor (Profile of Mood States, self-report measure).
  Depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University, Leiden, South Holland, Netherlands